CLINICAL TRIAL: NCT00503867
Title: A Pilot Study of Yttrium-90 Microspheres (SIR-Spheres®) Therapy for the Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: SIR-Spheres® for the Treatment of Unresectable Hepatocellular Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low patient recruitment
Sponsor: Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STX 0106
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Carcinoma, Hepatocellular; Hepatoma
Keywords: unresectable hepatocellular carcinoma; HCC; SIR-Spheres; Y-90 Microspheres; brachytherapy; Selective Internal Radiation Therapy (SIRT); liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SIR-Spheres microspheres (Experimental): SIR-Spheres microspheres
  Interventions: Device: SIR-Spheres microspheres

INTERVENTIONS:
Device: SIR-Spheres microspheres — SIR-Spheres Yttrium-90 microspheres

SUMMARY:
The main purpose of this study is to determine the safety and toxicity of treatment with SIR-Spheres® in patients with unresectable primary liver cancer or hepatocellular carcinoma (HCC). Other purposes of this study include assessment of the effect of treatment on overall survival, the length of time it takes for the disease to worsen, if and how the treatment affects the patient's quality of life, and if and how the cancer responds to the treatment.

DETAILED DESCRIPTION:
This study is a multi-institutional, non-randomized pilot study that aims to assess the safety and toxicity of hepatic arterial radioembolization using SIR-Spheres yttrium-90 microspheres (SIR-Spheres microspheres) in the treatment of patients with unresectable primary hepatocellular carcinoma (HCC). The study aims to recruit 40 patients over a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* must have a confirmed diagnosis of HCC.
* at least 18 years of age.
* must have a confirmed diagnosis of HCC either by histological confirmation or, in a subject who exhibits a vascular liver mass in the presence of radiographically apparent cirrhosis, an alpha-fetoprotein (AFP) level greater than 500 International Units/milliliter (UI/ml).
* must present HCC that is not amenable to surgical resection or immediate liver transplantation, or that is not optimally treatable with local ablative techniques such as radio-frequency ablation due to its size, extent or presence of cirrhosis.
* must present measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as greater than or equal to 10 mm with spiral CT scan or greater than or equal to 20 mm using conventional techniques (CT, MRI).
* must present with a whole-liver tumor burden of greater than or equal to 15% and less than or equal to 70%
* must have an Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less.
* must have normal organ and marrow function

Exclusion criteria:

Includes both the listed contraindications to SIR-Spheres® and the exclusion criteria specific to the setting of this investigational study:

* hepatic artery directed therapy within the previous 6 months.
* chemotherapy within the previous 4 weeks
* have not recovered from adverse events due to agents administered previously
* Prior external hepatic radiation therapy for HCC, more than two prior systemic chemotherapy regimes for HCC or any other concomitant therapy for HCC
* Currently receiving any other investigational agents for the treatment of their cancer.
* Any extra-hepatic metastases other than metastatic disease found in the lung, bone and/or abdominal lymph nodes that are not otherwise life limiting.
* Any other concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least five years.
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
* Any of the following contraindications to angiography and selective visceral catheterization:

  * Bleeding diathesis
  * Severe peripheral vascular disease
  * Portal hypertension with hepatofugal flow
* Female subjects who are pregnant or currently breastfeeding.
* Refusal or inability to use effective means of contraception in men or women of childbearing potential.
* Current enrollment in any other investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-07-18 (Actual); Primary Completion 2010-03-09 (Actual); Study Completion 2010-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Murthy, MD, Principal Investigator — M.D. Anderson Cancer Center; T. Clark Gamblin, MD, Principal Investigator — UPMC Liver Cancer Center
Locations (4):
- United States (4):
  - Thomas Jefferson University - Kimmel Cancer Center, Philadelphia, Pennsylvania
  - UPMC Liver Cancer Center, Pittsburgh, Pennsylvania
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Originally there was a plan to share the data with the Data Monitoring Committee, however the study was closed early due to lack of enrollment and the Data Monitoring Committee did not convene.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three medical centers in the US enrolled 10 patients from July 18, 2007 to March 9, 2010.
Groups:
- SIR-Spheres Microspheres: Radioembolization treatment with SIR-Spheres microspheres is administered within 28 days of enrollment into the study.
Period: Overall Study
Arm/Group | SIR-Spheres Microspheres
Started | 10
Completed | 8
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Hepatic Arterial Radioembolization SIR-Spheres Microspheres: SIR-Spheres microspheres
  SIR-Spheres microspheres: SIR-Spheres Yttrium-90 microspheres
Arm/Group | Hepatic Arterial Radioembolization SIR-Spheres Microspheres
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 68.0 [47.5 to 80.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
ECOG performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status
  Participants
    0 (full activity) | 8
    1 (ambulatory restricted) | 2
Previous chemotherapy [Count of Participants; unit: Participants] — 1 cycle Nexavar, 800 mg BID
  Participants
    Yes | 1
    No | 9
Previous radiotherapy [Count of Participants; unit: Participants]
  Yes | 1
  No | 9
Disease characteristics [Count of Participants; unit: Participants] — Hepatocellular carcinoma staging systems to determine prognosis included Okuda Staging, Cancer of the Liver Italian Program [CLIP]) & tumor node metastasis (TNM) classification. Higher grades/score classes correlate to poorer prognosis.
  Okuda classification include cancer-related variables and liver function variables (Grade 1 to 3).
  CLIP staging combines Child-Pugh score with tumour criteria: morphology, portal invasion, & alpha fetoprotein levels. (Stage 0 to 6).
  TNM staging describe size and/or extension of the primary tumor (Grade 1 to 4).
  Participants
    Okuda Stage 1 | 10
    CLIP score Class 1 | 4
    CLIP score Class 2 | 2
    CLIP score Class Unknown | 4
    Cirrhosis (Yes) | 8
    Cirrhosis (No) | 2
    TNM Classification of Primary Tumor, T2 | 2
    TNM Classification of Primary Tumor, T3 | 6
    TNM Classification of Primary Tumor, T4 | 2
    TNM Classification of regional lymph nodes (No) | 10
    Hepatitis B (Yes) | 1
    Hepatitis B (No) | 9
    Hepatitis C (Yes) | 3
    Hepatitis C (No) | 7
    Metabolic Liver Disease (No) | 10
    History of alcohol abuse (Yes) | 3
    History of alcohol abuse (No) | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Grade 3 or Higher
Description: Using the National Cancer Institute Common Terminology Criteria (NCI-CTC) version 3.0 as recorded in the case report form.
Time Frame: From date of enrollment until the date of death from any cause assessed up 24 weeks.
Population: Safety population - all patients who received initial SIRT treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SIR-Spheres Microspheres
Number analyzed (Participants) | 10
Participants | 3

2. Secondary Outcome: Time to Disease Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 52 weeks.
Population: This outcome measure was not assessed as no data was collected prior to termination of the study.
Arm/Group | SIR-Spheres Microspheres
Number analyzed (Participants) | 0

3. Secondary Outcome: Tumor Response Rate
Description: Tumour response rates estimated by the proportion of patients with a best response of CR, PR or SD by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) with corresponding exact 90% confidence limits being reported. Per RECIST v1.0 for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: as for outcome 2
Population: This outcome measure was not assessed as no data was collected prior to termination of the study.
Arm/Group | SIR-Spheres Microspheres
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Health-related Quality of Life
Time Frame: 52 weeks
Population: This outcome measure was not assessed as no data was collected prior to termination of the study.
Arm/Group | SIR-Spheres Microspheres
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time interval between the date of enrollment and the date of death from any cause.
Time Frame: as for outcome 2
Population: This outcome measure was not assessed as no data was collected prior to termination of the study.
Arm/Group | SIR-Spheres Microspheres
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From consent until 24 weeks post last dose of protocol chemotherapy.
Arm/Group | SIR-Spheres Microspheres
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIR-Spheres Microspheres (N=10)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
International Normalised Radio Increased (Investigations) | 1 (1)
Asthenia (General disorders) | 1 (1)
Dyspnoea (Cardiac disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Abdominal Distention (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No